CLINICAL TRIAL: NCT05246787
Title: The Effect of the Shotblocker and Breastfeeding on Pain and Comfort Level During Heel Lance Procedure in Newborns: Randomized Controlled Trial
Brief Title: Shotblocker and Breastfeeding on Pain/Comfort During Heel Lance
Acronym: heellance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BUCH 595
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Pain, Acute; Comfort
Keywords: breastfeeding; shotblocker
MeSH Terms: conditions — Acute Pain; Breast Feeding | interventions — Lactation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: attempt will be videotaped, outcome evaluators will be blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Breastfeeding intervention (Experimental): The baby will be placed on the mother's lap 2 minutes before the procedure. 2 minutes before the heel lance, the mother starts to breastfeed her baby and continues to breastfeed throughout the procedure and until the last touch to baby. If necessary, the researcher may verbally warn the mother in a calm tone to continue breastfeeding throughout the procedure. During the resting period (last 2 minutes) after the blood draw is completed, the baby stays on the mother's lap.
  Interventions: Behavioral: breastfeeding
- Shotblocker intervention (Experimental): 2 minutes before the procedure, the baby will be placed on the mother's lap. ShotBlocker is a small plastic tool that is blunt, short, has many points in contact with the skin, does not contain drugs, is in the shape of a horseshoe, invasive interventions can be applied through the space in the middle. It is positioned on the skin before the invasive procedure. The investigator should make sure that the contact points touch the skin. Shotblocker is pressed firmly for 20 seconds before the intervention, it is pulled from the area and the heel is pierced with the lancet. After Shotblocker is applied to the skin, invasive intervention should be performed within 30 seconds and the protocol should be followed. During the resting period (last 2 minutes) after the heel lance is completed, the baby stays on the mother's lap.
  Interventions: Device: shotblocker
- Breastfeeding and Shotblocker intervention (Experimental): The baby will be placed on the mother's lap 2 minutes before the procedure. 2 minutes before the heel lance, the mother starts to breastfeed her baby and continues to breastfeed throughout the procedure and until the last touch to baby. The investigator should make sure that the contact points touch the skin. Shotblocker is pressed firmly for 20 seconds before the intervention, it is pulled from the area and the heel is pierced with the lancet. After Shotblocker is applied to the skin, invasive intervention should be performed within 30 seconds and the protocol should be followed. During the resting period (last 2 minutes) after the heel lance is completed, the baby stays on the mother's lap.
  Interventions: Combination Product: Breastfeeding and Shotblocker
- Control group/ Standard Care (No Intervention): The baby is placed on the mother's lap 2 minutes before the procedure and the mother is provided to hold the baby effectively and graspingly. Standard heel lance procedure is applied. No additional interventions are applied to the baby. During the resting period (last 2 minutes) after the heel lance is completed, the baby stays on the mother's lap.

INTERVENTIONS:
Behavioral: breastfeeding — nonphamacological methods
  Arms: Breastfeeding intervention
Combination Product: Breastfeeding and Shotblocker — combined Breastfeeding and Shotblocker device
  Arms: Breastfeeding and Shotblocker intervention
Device: shotblocker — it is a small plastic tool
  Arms: Shotblocker intervention

SUMMARY:
Shotblocker and breastfeeding are an attempt to reduce pain during invasive procedures in newborns. This study was planned to evaluate the effect of non-pharmacological interventions on the pain and comfort level of newborns, whose heel blood will be taken in the 1st Level Neonatal Intensive Care Unit.

DETAILED DESCRIPTION:
Hypotheses H1: Newborns who undergo breastfeeding attempt during heel lance procedure feel less pain and have a higher comfort level.

H2: Newborns who undergo breastfeeding attempt and are applied shotblocker during heel lance procedure feel less pain and have a higher comfort level.

H3: Newborns who undergo shotblocker intervention during heel lance procedure feel less pain and have a higher comfort level.

H4: There are a difference between the comfort levels, HR and PO2 of newborns in terms of group, group-time and time according to the intervention applied.

Data collection process Mothers of newborns whose heel blood will be taken will be informed about the research. Consent will be obtained from the mother regarding the video recording during the heel lance precedure. After informed consent is obtained, it will be determined which group the newborn belongs to by stratified randomization.

A standard approach will be applied to all newborns. Standard approach involves performing the heel lance procedure on the caregiver's lap. Heel lance procedure will be scheduled between 09:00 and 10:00 in the morning, one hour after babies are breastfed. Babies to be included in the study in each group; they will be in their beds, in the undisturbed rest period, until 30 minutes before the start of the test. All babies; 2 minutes before, during and up to 2 minutes after blood collection; they will be video-recorded including their heart rate, faces, and upper and lower extremities (especially the heel to be operated). No additional care will be given to ensure physiological stability during each intervention (breastfeeding, shotblocker, etc.)

ELIGIBILITY:
Inclusion Criteria:

* Birth week is between 34-42 weeks,
* Postnatal in the first 10 days
* Birth weight is between 2500-4000 grams,
* Stable general condition,
* Being with her mother and literate,
* Breastfeeding,
* Newborns of mothers who agreed to participate in the study

Exclusion Criteria:

* In need of oxygen support,
* Unsuccessful heel lance attempt, patients whose heel lance cannot be taken in 30 sec.(in groups with shotblocker)
* Needing parenteral nutrition,
* Receiving analgesic treatment,
* Having physical, metabolic and genetic diseases,
* Having a mental or mental health problem in the mother
* Non-breastfed newborns
* Newborns hospitalized in the 3rd and 4th level neonatal intensive care unit

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | during the heel lance
  Turkish validity and reliability were established. Reliability values were found to be 0.83, 0.83, 0.86 before, during and after the procedure, respectively. Newborn infant pain scale is a likert-type scale consisting of 6 parameters, facial movements (0; relaxed, 1; restless), crying (0; no crying, 1; groaning, 2; loud crying), breathing (0; comfortable, 1; variable-irregular), arm (0: relaxed-free, 1; flexion-extension), leg (0; comfortable-free, 1; flexion-extension) and sleep-wake (0; sleeping-waking peaceful, 1; restless).
The Newborn Comfort Behavior Scale (NEAS) | during the heel lance
  The newborn comfort behavior scale is a Likert type scale developed to evaluate the comfort needs, pain and distress of newborn babies.his scale consists of six parameters: alertness, agitation, respiratory response/crying, body movements, facial tension and muscle tone.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, pHD, Principal Investigator — RN, PhD, Assoc. Prof.
Locations (2):
- Turkey (Türkiye) (2):
  - Gülçin Özalp Gerçeker, Izmir
  - Dr. Behçet Uz Children Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dinc C, Gerceker GO, Kalkanli O. The effect of the ShotBlocker(R) and breastfeeding on pain and comfort level during heel lance procedure in newborns: randomized controlled trial. Intensive Crit Care Nurs. 2025 Dec;91:104164. doi: 10.1016/j.iccn.2025.104164. Epub 2025 Jul 26. PMID 40716331